CLINICAL TRIAL: NCT00178776
Title: A Transtheoretical Model Group Therapy for Cocaine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Professor, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01DA015453-02 (NIH); R01DA015453-02 (NIH); UT CPHS ID - HSC-MS-02-138 (Other: University of Texas Health Science Center Houston)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2014-09

CONDITIONS: Cocaine Use Disorders
Keywords: Group; Therapy; Cocaine; Drugs; Trial; Outcome; Study; Feasibility; Transtheoretical; Stages; Motivation; Change
MeSH Terms: interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transtheoretical Model Group (Experimental)
  Interventions: Behavioral: Transtheoretical Model Group Therapy
- Education / Advice (Active Comparator)
  Interventions: Behavioral: Education & Advice

INTERVENTIONS:
Behavioral: Transtheoretical Model Group Therapy
  Arms: Transtheoretical Model Group
Behavioral: Education & Advice
  Arms: Education / Advice

SUMMARY:
The purpose of this study is to determine the feasibility and promise of a recently manualized group therapy based on the Transtheoretical Model for cocaine use disorders.

DETAILED DESCRIPTION:
Cocaine use in the general population is a significant and costly problem. Novel and innovative interventions targeting cocaine abuse are needed. The Transtheoretical Model of behavior change (TTM) offers a comprehensive framework for understanding, measuring, and intervening in behavior change and provides a strong theoretical foundation upon which effective treatments for substance abuse can be developed. The proposed Stage 1 research will pilot test a novel and innovative behavioral group therapy for cocaine users based on the TTM. In Phase 1, investigators will modify the newly developed Group Treatment for Substance Abuse: A Stages-of-Change Therapy Manual (Velasquez, Maurer, Crouch & DiClemente, 2001) to specifically target cocaine abuse resulting in a twelve-session, group intervention and accompanying therapy manual based on the TTM stages and processes of change: six "early stage" sessions targeting the experiential processes of change, and six "later stage" sessions targeting the behavioral processes of change. Phase 2 will consist of a pilot trial to evaluate the TTM group therapy with cocaine abusing patients. A randomized, controlled, between groups design will be used in which cocaine abusers (N=80) are assigned to one of two group treatment conditions: TTM therapy or Education/Advice. Participants will be recruited from Houston and surrounding communities through the Substance Abuse Research Center at the University of Texas Health Science Center Mental Sciences Institute. We expect the delivery of the TTM therapy for cocaine users to be feasible and acceptable, and to produce significant patient improvement. Cocaine outcomes will be assessed via objective (urine and drug analysis) and self-report measures. This Stage I research will contribute important theoretical and empirical information concerning the promise of a new and innovative intervention for cocaine abusers, and will provide the basis for a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: Male and female adults (ages 18-65 years old), of any race, who meet DSM-IV criteria for cocaine abuse or dependence disorder will be recruited. In addition, eligible participants must be:

* (1) judged to be in generally good physical and psychiatric health except for possible acute drug related problems;
* (2) willing and able to participate in the 6-week, group outpatient treatment;
* (3) able to provide the name of at least one person who can generally locate their whereabouts; and
* (4) willing to be followed for 3 months after treatment ends.

Potential subjects with simple drug charges whose legal contacts are willing to forego data revelation will be included. Although cocaine dependence will be the primary drug for which patients are seeking treatment, we will not exclude participants who are abusing additional substances.

Exclusion Criteria:

Individuals will be ineligible for study participation based on the following criteria:

* (1) current diagnosis of an Axis I psychiatric disorder other than cocaine dependence;
* (2) current psychiatric symptoms requiring medication;
* (3) severe medical, cognitive and /or psychiatric impairment that precludes cooperation with study protocol;
* (4) substance withdrawal symptoms requiring medical attention;
* (5) currently receiving other psychosocial therapy for substance abuse with the exception of AA, NA or CA;
* (6) impending incarceration;
* (7) inability to read, write, speak English;
* (8) inability or unwillingness to participate in the 6-week, group outpatient treatment (e.g., halfway house or other aftercare program restrictions).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2003-10; Primary Completion 2006-11 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Urinalysis indicating presence or absence of cocaine metabolites, used to calculate percent days abstinent, collected at intake, once weekly during the 6 week group treatment phase, at post-treatment, and 3 months.

SECONDARY OUTCOMES:
Secondary Outcome Measures Related to Cocaine and other Drug Use:
1) Timeline Follow-Back (self-reported use / percent days
abstinent)
2) Cocaine Craving Worksheet (self report)
3) Cocaine Negative Consequences Checklist (self report)
4) Addiction Severity Index (ASI; Interviewer Administered)
5) Blood Alcohol Breath (biological)
6) Substance Use Report (self report)
Secondary Outcome Measures Related to Feasibility of the Group Therapy:
1) Participation / Attendance / Retention
2) MI Scale (Therapist Adherence)
3) Treatment Satisfaction Questionnaire
4) Group Therapy Alliance Scale
5) Group Atmosphere Scale
6) Therapist Treatment Evaluation
Secondary Outcome Measures Related to Psychiatric Symptoms:
1) Beck Depression Inventory (BDI-II)
2) Brief Symptom Inventory (BSI)
Secondary Outcomes Related to Functioning:
1) HIV Knowledge Questionnaire
2) Risk Behavior Assessment
3) SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Mary Marden Velasquez, Ph.D., Principal Investigator — University of Texas Houston Medical School, Dept. of Family & Community Medicine
Locations (1):
- University of Texas Houston Mental Sciences Institute, Houston, Texas, United States

REFERENCES:
- [Background] Velasquez, M. M., Maurer, G. G., Crouch, C., & DiClemente, C. C. (2001). Group treatment for substance abuse: A stages-of-change therapy manual. New York: Guilford Press.